CLINICAL TRIAL: NCT02285790
Title: Treatment of Basal Cell Carcinoma Using a One-stop-shop With Reflectance Confocal Microscopy: a Randomized Controlled Multicenter Trial
Brief Title: One-stop-shop Study for Treatment of Basal Cell Carcinoma Using Reflectance Confocal Microscopy
Acronym: B-OSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: The Netherlands Cancer Institute (Other)
Responsible Party: Principal Investigator, Daniel Kadouch, Prof. dr. M.A. de Rie, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-OSS 2014_244
Record Dates: First submitted 2014-11-01; First posted 2014-11-07 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Carcinoma, Basal Cell
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — Microscopy, Confocal; Biopsy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RCM-OSS procedure (Experimental): The Vivascope 1500 will be used (CE certified, Lucid Technologies, Henrietta, NY, USA). Reflectance confocal microscopy (RCM) imaging will be performed for intended use only and interpreted on the Vivascope workstation by two investigators independently at both study locations. The investigators will be blinded to the results of the reference standard. After RCM imaging subjects will receive OSS surgical excision according to subtype. Clinically suspected primary BCCs that are not confirmed by RCM will also receive surgical treatment with a margin of 3mm.
  Interventions: Device: Reflectance confocal microscopy; Procedure: Surgical excision
- Standard of care procedure (Active Comparator): Clinical suspected primary BCCs, of all subtypes, will be diagnosed by conventional 3mm punch biopsy of the most elevated part of the lesion. Punch biopsies will be performed under local anesthetics using 1% xylocaine/adrenaline. HE stained sections of the punch biopsies will be evaluated by an experienced board certified pathologist. Subjects will receive surgical excision according to subtype within 6 weeks after punch biopsy has been performed. Clinically suspected new primary BCCs that are not confirmed by punch biopsy will also receive surgical treatment with a margin of 3mm.
  Interventions: Procedure: Punch biopsy; Procedure: Surgical excision

INTERVENTIONS:
Device: Reflectance confocal microscopy
  Other Names: Confocal microscopy; Vivascope 1500
  Arms: RCM-OSS procedure
Procedure: Punch biopsy
  Other Names: Biopsy
  Arms: Standard of care procedure
Procedure: Surgical excision — Excision of the suspected basal cell carcinoma lesion under local anesthetics
  Other Names: Surgical removal; Surgery

SUMMARY:
The purpose of this study is to assess the efficacy and safety of the one-stop-shop concept, using real-time in vivo reflectance confocal microscopy as diagnostic tool, prior to surgical management of new primary basal cell carcinoma

DETAILED DESCRIPTION:
Basal cell carcinoma (BCC) is the most common cancer diagnosed in white populations worldwide. The rising incidence of BCCs is becoming a major worldwide public health problem (1,11). Between 1973 and 2009, the European standardized rate quadrupled from 40 to 165 per 100,000 person-years for men and from 34 to 157 for women, most probably as a result of more intensive UV exposure (12). This is supported by previous published epidemiological literature indicating that ultraviolet radiation is an important risk factor for BCC with a significant increase among outdoor workers (13,14). Despite the low mortality from BCC, multiple and recurring tumors confer a high morbidity and considerable burden for health care providers and health budgets. Although BCC does not seem to have a high effect on patients' quality of life, patients suffering from BCC are definitely interested in efficacy, low recurrence rates and cosmetic outcome of their therapies.(15). Meanwhile resources available at hospitals have not increased proportionally and therefore optimizing effectiveness of present treatment modalities in daily dermatologic practice is mandatory (16).

Clinically, BCC are characterized by small, translucent, or pearly papules, with raised teleangiectatic edges (17) . Most of the BCC occur in sun-exposed skin of the head and neck area (18,19). Sensitivity and positive predictive value for the clinical diagnosing of BCC by dermatologists has been reported to be 95.4% and 85.9%, respectively (20). However, dividing between BCC subtypes is not always possible upon clinical assessment. To date, histological analysis of punch biopsy remains the golden standard to confirm the clinical diagnosis of BCCs and dividing between the following subtypes: nodular (nBCC), micronodular (mnBCC), infiltrating (iBCC) and superficial (sBCC) (10). Of those, nBCC and sBCC have a less aggressive growth pattern in comparison to mnBCC and iBCC. Additionally, mixed type BCC (mtBCC) can be defined as a combination of subtypes and are frequently composed of aggressive subtypes (21). Surgical excision remains the standard of treatment, with Mohs micrographic surgery typically utilized for high-risk lesions (22). Based upon the histological growth pattern, BCC are surgically removed with a margin of either 3mm (nBCC and sBCC) or 5mm (mnBCC, iBCC) in accordance with current Dutch guidelines (10).

Due to the rising incidence of BCC there is a need for more efficient, non-invasive methods to diagnose BCCs. The use of real-time in vivo reflectance confocal microscopy (RCM) to diagnose BCCs has proven successful to address this need. Various studies have demonstrated that RCM is safe and accurate (sensitivity and specificity) to diagnose BCCs(2-6). Reported sensitivity and specificity for RCM in diagnosing BCC range from 83%-100% and 79%-97%, respectively (7). Furthermore, Peppelman et al. and Longo et al. recently reported on RCM features that might divide between nodular, micronodular, superficial and infiltrative subtypes of BCC (8,9).

In 2012, van der Geer et al reported on the feasibility of a one-stop-shop (OSS) concept for the treatment of skin cancer patients (23). One-stop-shop implies that at the day of the initial outpatient clinic consultation, diagnosis and treatment plan both take place. In their study, pre-operative frozen section histology was used to confirm BCC diagnosis and subtype. The mean throughput time was 4 hours and 7 min, no complications were observed, and patient satisfaction was high (23). Incorporating RCM as non-invasive diagnostic tool in a BCC OSS concept for lesions suitable for conventional surgical excision might further reduce time between clinical diagnosis and treatment, administrative workload and costs.

The aim of our study is to assess the efficacy and safety of the one-stop-shop concept, using real-time in vivo reflectance confocal microscopy (Vivascope 1500; Lucid Technologies, Henrietta, NY, USA) as diagnostic tool, prior to surgical management of new primary BCCs, of all subtypes, in the general population.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically suspected new primary BCC as assessed by an experienced board certified dermatologist
* Patients seen at the outpatient clinic before 12h00 AM will be eligible to participate
* Patient is willing and able to give written informed consent
* BCC lesion is suitable for conventional surgical excision under local anesthetics
* BCC lesion is present since at least 1 month

Exclusion Criteria:

* BCC lesion in a high-risk location of the face (H-zone and ears)
* Contra-indication for conventional surgical excision (primary surgical closure seems not achievable)
* Recurrent BCC lesion (BCC that has been previously unsuccessfully treated) Macroscopic ulcerating BCC lesions (not feasible for RCM analysis due to technical reasons)
* Patients with basal cell nevus syndrome
* Patients treated with hedgehog inhibitor medication
* Patients with a history of hypersensitivity to and/ or a history of allergy to local anesthesia
* Unavailability within the following 6 weeks (for example due to holiday or sports)
* Patients not competent to understand the procedures involved

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-01; Primary Completion 2015-10 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Comparison between one stop shop using reflectance confocal microscopy in the surgical treatment of BCC and current standard of care using punch biopsy, by assessing incomplete surgical excision on the final pathology report. | Within the first week after surgical excision of suspected BCC lesion
  Assessment will be performed by an experienced board certified pathologist. The number of incomplete excisions will be compared between study- and control group.

SECONDARY OUTCOMES:
Comparison of the diagnostic accuracy (sensitivity and specificity) between RCM and punch biopsy in both diagnosing and subtyping BCCs | Within the first week after surgical excision of suspected BCC lesion
  Sensitivity and specificity of RCM for diagnosing and subtyping BCC, will be separately analyzed by comparing RCM diagnosis and subtype with final pathology reports of the study group. This will be performed by using unidentifiable saved RCM images of all included lesions of the study group.
Comparison of patient satisfaction between study group and standard of care (control) group by using a standardized web-based questionnaire for patient reported outcome in the management of skin diseases (www.huidvragen.info) | As assessed at the post-operative visit 3 months after surgical excision
  An adjusted version of this web-based questionnaire has previously been published to assess patient satisfaction among patients suffering from psoriasis (van Cranenburgh OD et al. Satisfaction with treatment among patients with psoriasis: a web-based survey study. Br J Dermatol. 2013 Aug;169(2):398-405). The outcome of the questionnaire will be compared between study- and control group.

OTHER OUTCOMES:
Comparison of throughput time, defined by the time between arrival at consultation until end of surgical treatment at our outpatient clinic, between study group and standard of care (control) group. | As assessed at the post-operative visit 3 months after surgical excision

CONTACTS AND LOCATIONS:
Overall Officials: Menno A. de Rie, MD, PhD, Principal Investigator — Head of Department
Locations (2):
- Netherlands (2):
  - Dutch Cancer Institute, Amsterdam, North Holland
  - Academic_Medical_Center, Amsterdam, North Holland

REFERENCES:
- [Background] Lomas A, Leonardi-Bee J, Bath-Hextall F. A systematic review of worldwide incidence of nonmelanoma skin cancer. Br J Dermatol. 2012 May;166(5):1069-80. doi: 10.1111/j.1365-2133.2012.10830.x. PMID 22251204
- [Background] Sauermann K, Gambichler T, Wilmert M, Rotterdam S, Stucker M, Altmeyer P, Hoffmann K. Investigation of basal cell carcinoma [correction of carcionoma] by confocal laser scanning microscopy in vivo. Skin Res Technol. 2002 Aug;8(3):141-7. doi: 10.1034/j.1600-0846.2002.20345.x. PMID 12236882
- [Background] Gonzalez S, Tannous Z. Real-time, in vivo confocal reflectance microscopy of basal cell carcinoma. J Am Acad Dermatol. 2002 Dec;47(6):869-74. doi: 10.1067/mjd.2002.124690. PMID 12451371
- [Background] van der Geer S, Reijers HA, van Tuijl HF, de Vries H, Krekels GA. Need for a new skin cancer management strategy. Arch Dermatol. 2010 Mar;146(3):332-6. doi: 10.1001/archdermatol.2010.1. PMID 20231509
- [Background] van der Geer S, Frunt M, Romero HL, Dellaert NP, Jansen-Vullers MH, Demeyere TB, Neumann HA, Krekels GA. One-stop-shop treatment for basal cell carcinoma, part of a new disease management strategy. J Eur Acad Dermatol Venereol. 2012 Sep;26(9):1154-7. doi: 10.1111/j.1468-3083.2011.04184.x. Epub 2011 Jul 19. PMID 21771105
- [Background] van Cranenburgh OD, de Korte J, Sprangers MA, de Rie MA, Smets EM. Satisfaction with treatment among patients with psoriasis: a web-based survey study. Br J Dermatol. 2013 Aug;169(2):398-405. doi: 10.1111/bjd.12372. PMID 23565643
- [Derived] Kadouch DJ, Wolkerstorfer A, Elshot Y, Zupan-Kajcovski B, Crijns MB, Starink MV, Bekkenk MW, van der Wal AC, Spuls PI, de Rie MA. Treatment of Basal Cell Carcinoma Using a One-Stop-Shop With Reflectance Confocal Microscopy: Study Design and Protocol of a Randomized Controlled Multicenter Trial. JMIR Res Protoc. 2015 Sep 10;4(3):e109. doi: 10.2196/resprot.4303. PMID 26362616
- See also: Kadouch et al., In vivo confocal microscopy of basal cell carcinoma: a systematic review of diagnostic accuracy. PROSPERO 2014:CRD42014010379 — http://www.crd.york.ac.uk/PROSPERO/display_record.asp?ID=CRD42014010379